CLINICAL TRIAL: NCT00732498
Title: Phase II Trial Of Yttrium-90-Ibritumomab Tiuxetan (Zevalin®) Radioimmunotherapy After Cytoreduction With ESHAP Chemotherapy In Patients With Relapsed Follicular Non-Hodgkin's Lymphoma
Brief Title: Rituximab, Yttrium Y 90 Ibritumomab Tiuxetan in Patients W/Relapsed Stage II, III, or IV Follicular NHL
Acronym: ESHAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-0303-04; P30CA023074 (NIH); CDR0000597508 (Other: PDQ #); 0500000303 (Other: UofA IRB #)
Record Dates: First submitted 2008-08-09; First posted 2008-08-12 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Etoposide; Cytarabine; Cisplatin; Rituximab; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ESHAP followed by Zevalin and Rituximab (Experimental): Etoposide, Methylprednisolone, Cytarabine, Cisplatin (ESHAP) infusion X 2 Cycles followed by Rituximab and In-Zevalin or Y-Zevalin.
  Interventions: Drug: Methylprednisolone; Drug: Etoposide; Drug: Cytarabine; Drug: Cisplatin; Drug: Rituximab; Drug: In-Zevalin; Drug: Y-Zevalin

INTERVENTIONS:
Drug: Methylprednisolone — 250 mg/m2/day IV over 1 hour days 1,2,3,4 every 28 days for 2 cycles. If bone marrow <25% involved and expected biodistribution after 2 cycles yttrium-90-ibritumomab tiuxetan (Zevalin) to be administered.
  Other Names: Methylprednisolone sodium succinate; Solu-Medrol
Drug: Etoposide — 40 mg/day IV over 1 hour days 1,2,3,4 every 28 days for 2 cycles. If bone marrow <25% involved and expected biodistribution after 2 cycles yttrium-90-ibritumomab tiuxetan (Zevalin) to be administered.
  Other Names: Vespesid
Drug: Cytarabine — 2000 mg/m2 IV over 2 hours days 4 every 28 days for 2 cycles. If bone marrow <25% involved and expected biodistribution after 2 cycles yttrium-90-ibritumomab tiuxetan (Zevalin) to be administered.
  Other Names: Cytosine Arabinoside
Drug: Cisplatin — 25 mg/m2/day IV at 1mg/min days 1,2,3,4 every 28 days for 2 cycles. If bone marrow <25% involved and expected biodistribution after 2 cycles yttrium-90-ibritumomab tiuxetan (Zevalin) to be administered.
  Other Names: CDDP
Drug: Rituximab — 250 mg/m2 slow IV over days 1, then 7,8 or 9 prior to In Zevalin. Rituximab + Zevalin regimen is given 4-6 weeks after completion of 2 cycles of ESHAP. Treatment can be completed within 7-9 days in an outpatient setting.
  Other Names: Ibritumomab; Rituxan
Drug: In-Zevalin — 5 mCi slow IV push over 10 minutes days 1. Given within 4 hours after Rituximab.
  Other Names: Zevalin, Yttrium-90-Ibritumomab Tiuxetan
Drug: Y-Zevalin — Platelet counts from 100,000/mm3 to 149,000/mm3 will receive 0.3 mCi/kg. Platelet counts from >/= 150,000/mm3 will receive 0.4 mCi/kg, not to exceed 32 mCi Y Zevalin. Slow IV push over 10 minutes, days 7,8 or 9 given within 4 hours after Rituximab.
  Other Names: Yttrium-90-Ibritumomab Tiuxetan, Zevalin

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Radiolabeled monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Giving combination chemotherapy together with rituximab and yttrium Y 90 ibritumomab tiuxetan may kill more cancer cells.

PURPOSE: This phase II trial is studying giving combination chemotherapy followed by rituximab and yttrium Y 90 ibritumomab tiuxetan to see how well it works in treating patients with relapsed stage II, stage III, or stage IV follicular non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the 1-year progression-free survival of patients with relapsed stage II-IV follicular non-Hodgkin lymphoma treated with ESHAP chemotherapy for cytoreduction followed by yttrium Y 90 ibritumomab tiuxetan radioimmunotherapy.
* To evaluate the median time to progression in these patients.

Secondary

* To evaluate the overall and complete response rates in patients treated with this regimen.

OUTLINE:

* ESHAP chemotherapy: Patients receive ESHAP chemotherapy comprising etoposide IV over 1 hour, methylprednisolone IV, cisplatin IV on days 1-4, and cytarabine IV over 2 hours on day 1. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.
* Radioimmunotherapy: Between 4-6 weeks after completion of ESHAP chemotherapy, patients receive rituximab IV followed by indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1. Patients with < 25% bone marrow involvement and expected biodistribution proceed to treatment. Patients receive rituximab IV followed by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 7, 8, or 9.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of follicular non-Hodgkin lymphoma (NHL)
* Bulky stage II, stage III, or stage IV disease, Bulky disease is defined as any tumor measuring 10.0 cm or more or occupying ≥ one-third of the chest diameter
* In first, second, third, or fourth relapse after chemotherapy
* Unilateral or bilateral bone marrow aspirate and biopsy with cytogenetics within the past 42 days
* Tumor CD20 positive by either flow cytometry or immunoperoxidase staining of paraffin sections using anti-CD20 antibodies
* Bidimensionally measurable disease
* Patients with non-measurable disease in addition to measurable disease must have all non-measurable disease assessed within the past 42 days
* No presence of CNS lymphoma
* No chronic lymphocytic leukemia
* No HIV- or AIDS-related lymphoma
* No presence of pleural effusion
* Zubrod performance status 0-2
* ANC ≥ 1,500/μL (unless decreased counts are due to marrow involvement with NHL)
* Platelet count > 100,000/μL (unless decreased counts are due to marrow involvement with NHL)
* Serum creatinine ≤ 2.0 mg/dL
* Creatinine clearance ≤ 50 mL/min
* Serum bilirubin ≤ 2.0 mg/dL
* No renal insufficiency or renal failure
* No known HIV positivity
* Not pregnant or nursing
* No prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer with 5-year disease-free status
* No impaired bone marrow reserve, including any of the following:
* Hypocellular bone marrow (cellularity ≤ 15%)
* Marked ( ≥ 10%) reduction in bone marrow precursors of one or more cell lines (granulocytic, megakaryocytic, erythroid) (beyond that which would be expected for the patient's age and bone marrow cellularity)
* History of failed stem cell collection
* No serious, non-malignant disease or infection which, in the opinion of the investigator and/or sponsor, would compromise other protocol objectives
* At least 3 weeks since all prior therapy (6 weeks for rituximab) and recovered
* No prior myeloablative therapies with autologous bone marrow transplantation or peripheral blood stem cell rescue
* No prior radioimmunotherapy
* No prior external beam radiotherapy to > 25% of active bone marrow (involved field or regional)
* More than 4 weeks since prior major surgery, other than diagnostic surgery

Exclusion Criteria

Patients with impaired bone marrow reserve, as indicated by one or more of the following:

* Platelet count < 100,000 cells/mm3
* Hypocellular bone marrow (cellularity < or = 10%)
* Marked (> 10%) reduction in bone marrow precursors of one or more cell lines (granulocytic, megakaryocytic, erythroid) (beyond that which would be expected for the patient's age and bone marrow cellularity
* History of failed stem cell collection

Prior radioimmunotherapy

Presence of CNS lymphoma. Patients must not have clinical evidence of central nervous system (CNS) involvement by lymphoma.

Patients with abnormal liver function: total bilirubin > 2.0 mg/dL

Patients with abnormal renal function: serum creatinine > 2.0 mg/dL or creatinine clearance < 50 ml/min.

Patients who have received prior external beam radiation therapy to > 25% of active bone marrow (involved field or regional)

Patients who have received G-CSF or GM-CSF therapy within 2 weeks prior to treatment

Serious nonmalignant disease or infection which, in the opinion of the investigator and/or the sponsor, would compromise other protocol objectives

Major surgery, other than diagnostic surgery, within 4 weeks

Patients with pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-05-15 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O. Persky, MD, Principal Investigator — University of Arizona
Locations (1):
- The University of Arizona Cancer Center, Tucson, Arizona, United States

REFERENCES:
- See also: Journal Article — https://www.ncbi.nlm.nih.gov/pubmed/29471300

RESULTS

PARTICIPANT FLOW:
Groups:
- ESHAP Followed by Zevalin and Rituximab: Etoposide, Methylprednisolone, Cytarabine, Cisplatin (ESHAP) infusion X 2 Cycles followed by Rituximab and In-Zevalin or Y-Zevalin.
  Methylprednisolone: 250 mg/m2/day IV over 1 hour days 1,2,3,4 every 28 days for 2 cycles. If bone marrow <25% involved and expected biodistribution after 2 cycles yttrium-90-ibritumomab tiuxetan (Zevalin) to be administered.
  Etoposide: 40 mg/day IV over 1 hour days 1,2,3,4 every 28 days for 2 cycles. If bone marrow <25% involved and expected biodistribution after 2 cycles yttrium-90-ibritumomab tiuxetan (Zevalin) to be administered.
  Cytarabine: 2000 mg/m2 IV over 2 hours days 4 every 28 days for 2 cycles. If bone marrow <25% involved and expected biodistribution after 2 cycles yttrium-90-ibritumomab tiuxetan (Zevalin) to be administered.
  Cisplatin: 25 mg/m2/day IV at 1mg/min days 1,2,3,4 every 28 days for 2 cycles. If bone marrow <25% involved and expected biodistribution after 2 cycles yttrium-90-ibritumomab tiuxetan (Zevalin) to be admin
Period: Overall Study
Arm/Group | ESHAP Followed by Zevalin and Rituximab
Started | 28
Completed | 22
Not Completed | 6
Not completed — Ineligible | 1
Not completed — Adverse Event | 2
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | ESHAP Followed by Zevalin and Rituximab
Number analyzed (Participants) | 28
Age, Customized [Median (Standard Deviation); unit: years]
  Median age, years | 61 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 27
  Hispanic | 3
Region of Enrollment [Number; unit: participants]
  United States | 28
Baseline B Symptoms [Count of Participants; unit: Participants] — B symptoms refer to systemic symptoms of fever, night sweats, and weight loss.
  Participants | 15
Bone marrow involvement [Count of Participants; unit: Participants] | 12
Prior transplant history [Count of Participants; unit: Participants] | 1
Tumor bulk >5cm [Count of Participants; unit: Participants] | 7
Prior chemotherapy regimens [Count of Participants; unit: Participants]
  Zero cycles | 0
  One cycle | 16
  Two cycles | 7
  Three cycles | 3
  Four cycles | 2
Elevated beta2-microglobin [Count of Participants; unit: Participants] | 11
Follicular Lymphoma International Prognostic Index (FLIPI) [Count of Participants; unit: Participants] — Estimates overall survival based on clinical information. Measures survival from diagnosis.A FLIPI score of 0 to 1 is considered "low risk" with a 10 year overall survival of 70%. A score of 2 is considered "intermediate risk" with a 10 year overall survival of 50%. Finally, a score of ≥ 3 is considered "high risk" with a 10 year overall survival of 35%.
  Participants
    0 | 1
    1 | 4
    2 | 10
    3 | 8
    4 | 5
The Follicular Lymphoma International Prognostic Index-2 (FLIPI2) [Count of Participants; unit: Participants] — Estimates overall survival based on clinical information. FLIPI2 is applied at the time of treatment for follicular lymphoma.
  Participants
    0 | 4
    1 | 9
    2 | 8
    3 | 5
    4 | 2
Response to prior chemotherapy regimens [Count of Participants; unit: Participants]
  Complete reponse | 9
  Partial response | 4
  Stable disease | 1
  Progressive disease | 11
  Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 1 Year
Description: To evaluate the 1-year progression-free survival (PFS) of patients with relapsed follicular non-Hodgkin's lymphoma (NHL) treated with ESHAP chemotherapy for cytoreduction (2 cycles) followed by Ibritumomab tiuxetan (Zevalin) radioimmunotherapy.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | ESHAP Followed by Zevalin and Rituximab
Number analyzed (Participants) | 22
percentage of participants | 38

2. Primary Outcome: Median Time to Progression
Description: To evaluate the median TTP of patients with relapsed follicular NHL treated with ESHAP chemotherapy for cytoreduction (2 cycles) followed by Ibritumomab tiuxetan (Zevalin) radioimmunotherapy.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ESHAP Followed by Zevalin and Rituximab
Number analyzed (Participants) | 22
months | 10 [8.0 to 18.0]

3. Secondary Outcome: Overall Response Rate
Description: To evaluate the overall (ORR) response rate with relapsed follicular NHL treated with ESHAP chemotherapy for cytoreduction (2 cycles) followed by Ibritumomab tiuxetan (Zevalin) radioimmunotherapy. Descriptive and summary statistics for demographic and clinical variables obtained. The incidences of reported adverse events (AEs) tabulated. Kaplan-Meier survival analysis for PFS and OS performed on TPP. All the analyses were performed using Stata [12].
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | ESHAP Followed by Zevalin and Rituximab
Number analyzed (Participants) | 22
percentage of participants | 77.3

4. Secondary Outcome: Complete Response Rate
Description: To evaluate the complete (CR) response rate with relapsed follicular NHL treated with ESHAP chemotherapy for cytoreduction (2 cycles) followed by Ibritumomab tiuxetan (Zevalin) radioimmunotherapy
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | ESHAP Followed by Zevalin and Rituximab
Number analyzed (Participants) | 22
Participants | 10

ADVERSE EVENTS:
Time Frame: Five years
Arm/Group | ESHAP Followed by Zevalin and Rituximab
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 6/28
Other Adverse Events (participants affected / at risk) | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ESHAP Followed by Zevalin and Rituximab (N=28)
Perforated duodenal ulcer (Gastrointestinal disorders) | 1
Nausea/Vomiting (Gastrointestinal disorders) | 1
Myelodysplastic syndrome (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Metachronous colon carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ESHAP Followed by Zevalin and Rituximab (N=28)
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Fatigue (General disorders) | 21
Anemia (Blood and lymphatic system disorders) | 21
Leukopenia (Blood and lymphatic system disorders) | 19
Nausea (Gastrointestinal disorders) | 18
Pain (General disorders) | 16
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 9
Constipation (Gastrointestinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Dizziness (Nervous system disorders) | 6
Diarrhea (Gastrointestinal disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 4
Neuropathy (Nervous system disorders) | 5
Weight loss (Metabolism and nutrition disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Tinnitus (Ear and labyrinth disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT00732498/Prot_SAP_000.pdf